CLINICAL TRIAL: NCT06135701
Title: Femoral Artery Blood Flow During Rest and One-leg Knee Extensor Exercise in Patients With COPD
Acronym: COPD-DOPPLER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Milan Mohammad, BSc(Med) and principal investigator at Center for Aktiv Sundhed (CFAS), Rigshospitalet., Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-23049997
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: COPD; Healthy; Chronic Obstructive Pulmonary Disease
Keywords: Ultrasound; COPD; Test-retest
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Experimental setup Femoral blood flow will be measured by Doppler ultrasound at rest and during one-knee leg extensor exercise.
  Preliminary maximal knee extensor test The maximal workload (WLpeak) of the thigh muscles during one-legged knee-extensor exercise on a customized one-leg kicking chair will be determined.
  One-legged knee-extensor exercise protocol In rest upright and supine 0 watt 20%watt max 10 watt. This study day will be repeated within 2-7 days.
  Doppler ultrasound Doppler-based blood flow in the common femoral artery (QDop) is obtained using a linear probe (4.3-5.0 MHz) to obtain two-dimensional (2D) femoral arterial cross-sectional area (A) and mean blood velocity (v ̅).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD-patients (Experimental): The participants will be instructed to abstain from caffeine, nicotine, alcohol, and strenuous exercise all known to affect blood flow to the limb for 12 hours prior to the study day. After being placed on the one-leg kicking chair, baseline measurements will be performed, followed by passive leg movement for 2 minutes. Then participants will perform one-legged knee-extension exercise at submaximal intensity, first at 10% and then at 20% of the previously measured WLpeak, remaining 3.5 minutes at each level, while femoral blood flow is measured. This study day will be repeated within 2-10 days.
  Interventions: Diagnostic Test: One-legged knee-extensor exercise with Doppler measurements
- Matched healthy volunteers (Experimental): The participants will be instructed to abstain from caffeine, nicotine, alcohol, and strenuous exercise all known to affect blood flow to the limb for 12 hours prior to the study day. After being placed on the one-leg kicking chair, baseline measurements will be performed, followed by passive leg movement for 2 minutes. Then participants will perform one-legged knee-extension exercise at submaximal intensity, first at 10% and then at 20% of the previously measured WLpeak, remaining 3.5 minutes at each level, while femoral blood flow is measured. This study day will be repeated within 2-10 days.
  Interventions: Diagnostic Test: One-legged knee-extensor exercise with Doppler measurements

INTERVENTIONS:
Diagnostic Test: One-legged knee-extensor exercise with Doppler measurements — Doppler ultrasound is used while participants exercise according to the one-legged knee-extensor exercise model

SUMMARY:
Doppler ultrasound is generally considered to provide reliable femoral blood flow measurements between rest and exercise, and the blood flow response to exercise is widely believed to be reduced in patients with chronic obstructive pulmonary disease (COPD). However, the test-retest reliability of the method during one-leg knee extensor exercise has not previously been compared between matched healthy individuals.

DETAILED DESCRIPTION:
Experimental assessments of changes in skeletal muscle blood flow during exercise in humans are important for elucidating the factors that limit exercise capacity and adaptations, both in healthy humans, including athletes, as well as in various disease states with functional impairment, such as chronic obstructive pulmonary disease COPD). A classical 'gold standard' for measuring blood flow is thermodilution, and this has notably applied to provide data on femoral blood flow during exercise. Because thermodilution required invasive catheterization, many have replaced it with Doppler ultrasound, but the test-retest reliability of Doppler ultrasound in this context is unknown. However, many studies have used Doppler ultrasound to document that the femoral blood flow response to exercise is impaired in COPD, which ultimately affects oxygen uptake and thus exercise capacity, but the interpretation of these findings is currently hampered by the lack of knowledge regarding the test-retest reliability of the method in this patient group.

The investigators aim is to compare the femoral blood flow response to one-legged knee extensor exercise in patients with COPD vs. healthy participants, and to provide an estimate of the test-retest reliability the femoral blood flow measurements obtained by Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria for COPD patients:

* Men and women
* 45-80 years
* COPD (GOLD stage I to III)
* Forced expiratory volume in 1 sec (FEV1)/forced vital capacity ratio (FVC) < 0.8, FEV1 < 90% of predicted value
* Modified Medical Research Council score (mMRC 0 - 3) Resting arterial oxygenation > 90%

Exclusion Criteria for COPD patients:

* Symptoms of ischaemic heart disease
* Known heart failure
* Claudication
* Symptoms of disease within 2 weeks prior to the study
* Participation in pulmonary rehabilitation within 6 months
* Known malignant disease
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Inclusion Criteria for healthy matched controls:

* Men and women
* 45-80 years
* Normal FEV1, FVC, FEV1/FVC, and single-breath diffusion capacity
* Same sex, age (± 3 years) as the COPD patients

Exclusion Criteria for healthy matched controls:

* Known chronic lung disease
* Known ischaemic heart disease
* Known heart failure
* Symptoms of disease within 2 weeks prior to the study
* Known malignant disease
* Claudication
* Pregnancy
* Unstable cardiac arrhythmic disease
* Renal or liver dysfunction

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Between-day smallest real difference (SRD) for femoral blood flow at rest and at each relative exercise intensity in COPD vs. healthy controls | Measured at day 1 and day 2
  Doppler ultrasound measured blood flow during one leg knee extensor exercise with different intensities.
• Between-day coefficient of variance (CV) for femoral blood flow at rest and at each relative exercise intensity in COPD vs. healthy controls (co-primary) | Measured at day 1 and day 2
  Doppler ultrasound measured blood flow during one leg knee extensor exercise with different intensities.

SECONDARY OUTCOMES:
Femoral blood flow response to exercise at each relative exercise intensity in COPD vs. healthy controls (key secondary) | Measured at day 1 and day 2
  Doppler ultrasound measured blood flow during one leg knee extensor exercise with different intensities.
Between-day smallest real difference (SRD) for femoral blood flow at rest and at each absolute exercise intensity in COPD vs. healthy controls | Measured at day 1 and day 2
  Doppler ultrasound measured blood flow during one leg knee extensor exercise with different intensities.
• Between-day coefficient of variance (CV) for femoral blood flow at rest and at each absolute exercise intensity in COPD vs. healthy controls (co-primary) | Measured at day 1 and day 2
  Doppler ultrasound measured blood flow during one leg knee extensor exercise with different intensities.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Aktiv Sundhed (CFAS), Rigshospitalet, Copenhagen, Denmark., Copenhagen, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Can be retrieved upon request from primary investigator.